CLINICAL TRIAL: NCT02436304
Title: Safety and Efficacy of EXE844 Otic Suspension in the Treatment of Otitis Media at Time of Tympanostomy Tube Insertion
Brief Title: Safety and Efficacy of EXE844 Otic Suspension in Otitis Media at Time of Tympanostomy Tube Insertion (OMTT) - Study 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXE844b-C002
Record Dates: First submitted 2015-05-04; First posted 2015-05-06 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-07

CONDITIONS: Otitis Media With Effusion in Children; Otitis Media Recurrent
MeSH Terms: interventions — Middle Ear Ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EXE844 for 7 Days + Tubes (Experimental): EXE844 Sterile Otic Suspension, 0.3%, ototopical, 4 drops, twice daily (BID) in each ear for 7 days after Tympanostomy Tube Insertion
  Interventions: Drug: EXE844 Sterile Otic Suspension, 0.3%; Procedure: Tympanostomy Tube Insertion
- EXE844 for 3 Days + Tubes (Experimental): EXE844 Sterile Otic Suspension, 0.3%, ototopical, 4 drops BID in each ear for 3 days after Tympanostomy Tube Insertion
  Interventions: Drug: EXE844 Sterile Otic Suspension, 0.3%; Procedure: Tympanostomy Tube Insertion
- Tubes Only (Active Comparator): Bilateral myringotomy and tympanostomy tube insertion
  Interventions: Procedure: Tympanostomy Tube Insertion

INTERVENTIONS:
Drug: EXE844 Sterile Otic Suspension, 0.3%
  Arms: EXE844 for 3 Days + Tubes; EXE844 for 7 Days + Tubes
Procedure: Tympanostomy Tube Insertion — Surgical procedure for treating pediatric cases of recurrent or chronic otitis media

SUMMARY:
The purpose of this study is to evaluate EXE844 plus tympanostomy tubes compared to tympanostomy tubes only based on sustained clinical cure at end-of-therapy (EOT).

ELIGIBILITY:
Inclusion Criteria:

* Recurrent acute otitis media (RAOM) or chronic otitis media with effusion (COME) and eligible for bilateral myringotomy and tympanostomy tube insertion.
* Suspected bacterial infection at time of surgery in at least 1 ear.
* Willing to refrain from water immersion of the ears following surgery without the use of adequate ear protection during swimming, bathing, showering and other water-related activities.
* Legally Authorized Representative (LAR) must read and sign the informed consent.
* Parent or caregiver must agree to comply with the requirements of the study and administer study medication as directed, complete required study visits, and comply with the protocol.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Previous otologic or otologic-related surgery within the past 30 days or ongoing complications.
* Middle ear pathology in either ear other than otitis media.
* Current acute otitis externa (AOE), malignant otitis externa (MOE) or other conditions which could interfere with evaluation of the study drug.
* Any systemic disease or disorder, complicating factor or structural abnormality that would negatively affect the conduct or outcome of the study based upon assessment by the Investigator.
* Known or suspected allergy or hypersensitivity to quinolones or other active or inactive ingredients present in the medications to be used in the study.
* Other protocol-specified exclusion criteria may apply.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 404 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Ophtha-GCRA, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 19 study centers located in Canada (3) and the US (16).
Pre-assignment Details: Of the 404 enrolled, 48 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants (356).
Groups:
- EXE844 7 Days: EXE844 Sterile Otic Suspension, 0.3%, ototopical, 4 drops, twice daily (BID) in each ear for 7 days after Tympanostomy Tube Insertion
- EXE844 3 Days: EXE844 Sterile Otic Suspension, 0.3%, ototopical, 4 drops BID in each ear for 3 days after Tympanostomy Tube Insertion
Period: Overall Study
Arm/Group | EXE844 7 Days | EXE844 3 Days | Tubes Only
Started | 153 | 102 | 101
Completed | 153 | 100 | 100
Not Completed | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Randomized in error didn't meet I/E crit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants, including those who underwent concurrent adenoidectomy and/or tonsillectomy (Intent-to-treat (ITT) analysis set)
Groups:
- EXE844 7 Days: EXE844 Sterile Otic Suspension, 0.3%, ototopical, 4 drops, BID in each ear for 7 days after Tympanostomy Tube Insertion
- Total: Total of all reporting groups
Arm/Group | EXE844 7 Days | EXE844 3 Days | Tubes Only | Total
Number analyzed (Participants) | 153 | 102 | 101 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.3 (2.05) | 2.8 (2.31) | 2.6 (2.31) | 2.5 (2.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 43 | 40 | 136
  Male | 100 | 59 | 61 | 220

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Sustained Clinical Cure at Day 8
Description: Sustained clinical cure was defined as the absence of otorrhea in the study ear at Day 8 (end of treatment (EOT)) per the Investigator assessment. Participants were considered a treatment failure if, at any time during the course of the study, an alternative therapy was initiated to treat the post-surgical infection. All participants who had missing or indeterminate outcomes were considered a failure (same as baseline observation carried forward).
Time Frame: Day 8
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | EXE844 7 Days | EXE844 3 Days | Tubes Only
Number analyzed (Participants) | 153 | 102 | 101
percentage of participants | 77.1 | 75.5 | 65.3

2. Secondary Outcome: Percentage of Subjects With Microbiological Success at Day 14
Description: Microbiological success was attained if all pretherapy bacteria were absent in the study ear for the test-of-cure (TOC) specimen, which was presumed a success for subjects with no otorrhea at Day 14. Participants were considered a treatment failure if, at any time during the course of the study, an alternative therapy was initiated to treat the post-surgical infection. All participants who had missing or indeterminate outcomes were considered a failure (same as baseline observation carried forward).
Time Frame: Day 14
Population: This analysis population includes all ITT participants who were culture-positive at Day 1 in at least 1 ear (Microbiological Intent-to-Treat (MITT) analysis set)
Measure: Number; unit: percentage of participants
Arm/Group | EXE844 7 Days | EXE844 3 Days | Tubes Only
Number analyzed (Participants) | 80 | 58 | 52
percentage of participants | 72.5 | 69.0 | 51.9

3. Secondary Outcome: Time to Cessation of Otorrhea
Description: The time to cessation of otorrhea in the enrolled ear(s) was calculated as the number of days from the day of surgery to the absence of otorrhea (ie, no discharge) as reported by the parent/caregiver. Participants were considered a treatment failure if, at any time during the course of the study, an alternative therapy was initiated to treat the post-surgical infection. All participants who had missing or indeterminate outcomes were considered a failure (same as baseline observation carried forward).
Time Frame: Up to Day 14
Population: ITT analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | EXE844 7 Days | EXE844 3 Days | Tubes Only
Number analyzed (Participants) | 153 | 102 | 101
days | 2.5 [1.5 to 3.0] | 2.0 [1.0 to 3.0] | 1.5 [0.5 to 3.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 28 days). AEs are reported as pretreatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained as solicited comments from the study participants and as observations by the Investigator as outlined in the study protocol.
Groups:
- Pretreatment: All who consented to participate in the study prior to randomization
- EXE844 7 Days: All participants exposed to EXE844 Sterile Otic Suspension, 0.3% for 7 days after Tympanostomy Tube Insertion
- EXE844 3 Days: All participants exposed to EXE844 Sterile Otic Suspension, 0.3%, for 3 days after Tympanostomy Tube Insertion
- Tubes Only: All participants who underwent bilateral myringotomy and tympanostomy tube insertion only
Arm/Group | Pretreatment | EXE844 7 Days | EXE844 3 Days | Tubes Only
All-Cause Mortality (participants affected / at risk) | 0/404 | 0/153 | 0/102 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/404 | 0/153 | 0/102 | 0/101
Other Adverse Events (participants affected / at risk) | 2/404 | 39/153 | 19/102 | 13/101
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=404) | EXE844 7 Days (N=153) | EXE844 3 Days (N=102) | Tubes Only (N=101)
Ear Pain (Ear and labyrinth disorders) | 0 | 11 | 5 | 5
Pyrexia (General disorders) | 1 | 12 | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 10 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 6 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.